CLINICAL TRIAL: NCT01126242
Title: Tape Versus Semirigid Versus Lace-up Ankle Support in the Treatment of Acute Lateral Ankle Ligament Injury.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gelre Hospitals (Other)
Responsible Party: Principal Investigator, Michel P. J. van den Bekerom, MD, Gelre Hospitals
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-142
Record Dates: First submitted 2010-05-18; First posted 2010-05-19 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2010-04

CONDITIONS: Grade II and III Acute Lateral Ankle Ligament Injuries
Keywords: Ankle; ligament injuries; non-surgical treatment; tape; brace; orthotic device; bandage; cost-effectiveness; randomized trial
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- tape (Experimental): Group I will be treated with non-elastic adhesive tape around the affected ankle, applied by the 'van Unen-technique'. This technique is an alternative for the 'Coumans- technique'. The rationale of taping is to take the load off the injured tissue, to correct the biomechanics, to protect the injured part and to enhance proprioception and awareness of the injured tissue. Different materials can be used alone or in combination. The bandage material must have an adhesive layer which allows it to adhere to the skin and to itself. Since the direct stabilizing effect of a bandage lasts no longer than about half an hour, the positive effect is presumed to occur primarily through traction on the skin which stimulates muscular activity. Taping is a treatment that involves no loss of time, requires no crutches and is not attended with any ultimate impairment of function.
  Interventions: Device: Tape; Device: Semi rigid brace; Device: Lace-up brace
- Lace-up brace (Active Comparator): The ASO (Ankle Stabilizing Orthosis) fits into an athletic or street shoe. The ASO is made of thin, durable ballistic nylon - the same protective material used by law enforcement and military personnel. Support is achieved through exclusive non-stretch nylon stabilizing straps that mirror the stirrup technique of an athletic taping application. The calcaneus is captured, effectively locking the heel. The ASO ankle brace holds the ankle in a biomechanical neutral position, reducing either inversion or eversion type injuries or re-injuries.
  Interventions: Device: Tape; Device: Semi rigid brace; Device: Lace-up brace
- Semi rigid brace (Active Comparator): A semi-rigid brace, the M-step® from Medi®, will be applied. The foam gel in the pads continuously adapts to give an uninterrupted optimal fit to the constantly changing anatomical conditions, which therefore ensures a uniform compression. The ability of the foam gel pad to adapt allows one orthosis to be used for both the left and the right ankle. The pads are very light and have a soft fleecy surface. Even the edges of the outer moldings are generously padded. The M-step ankle orthosis can be quickly and securely applied by means of two Velcro fasteners; the Velcro fasteners can be detached from the outer shells and fixed individually.
  Interventions: Device: Tape; Device: Semi rigid brace; Device: Lace-up brace

INTERVENTIONS:
Device: Tape — Group I will be treated with non-elastic adhesive tape (Leukotape® Classic) around the affected ankle, applied by the 'van Unen-technique'.18 This technique is an alternative for the 'Coumans- technique'.15 The rationale of taping is to take the load off the injured tissue, to correct the biomechanics, to protect the injured part and to enhance proprioception and awareness of the injured tissue. Different materials can be used alone or in combination. The bandage material must have an adhesive layer which allows it to adhere to the skin and to itself. Since the direct stabilizing effect of a bandage lasts no longer than about half an hour, the positive effect is presumed to occur primarily through traction on the skin which stimulates muscular activity.
Device: Semi rigid brace — Group II will be treated by application of a semi-rigid brace, the M-step® from Medi®. The foam gel in the pads continuously adapts to give an uninterrupted optimal fit to the constantly changing anatomical conditions, which therefore ensures a uniform compression. The ability of the foam gel pad to adapt allows one orthosis to be used for both the left and the right ankle. The pads are very light and have a soft fleecy surface. Even the edges of the outer moldings are generously padded. The M-step ankle orthosis can be quickly and securely applied by means of two Velcro fasteners; the Velcro fasteners can be detached from the outer shells and fixed individually.
Device: Lace-up brace — Group III will be treated by application of a lace-up brace, the ASO brace. The ASO (Ankle Stabilizing Orthosis) fits into an athletic or street shoe. The ASO is made of thin, durable ballistic nylon - the same protective material used by law enforcement and military personnel. Support is achieved through exclusive non-stretch nylon stabilizing straps that mirror the stirrup technique of an athletic taping application. The calcaneus is captured, effectively locking the heel. The ASO ankle brace holds the ankle in a biomechanical neutral position, reducing either inversion or eversion type injuries or re-injuries.

SUMMARY:
The objective of this study is to compare tape versus semi rigid support versus lace up brace treatment for acute lateral ankle ligament injuries with regard to clinical outcome and cost effectiveness.

There is a difference of 10 in functional outcome (Karlsson Score) between non-elastic adhesive taping and semi-rigid and lace-up ankle support, in favour of the last, for the treatment of acute lateral ankle ligament injury at 6 months follow-up.

DETAILED DESCRIPTION:
This study is designed as a single blind prospective randomized controlled trial to evaluate the difference in functional outcome after treatment with tape versus semi-rigid versus lace-up ankle support (brace) for grade II and III acute lateral ankle ligament injuries. The patients will be randomly allocated into one of the three groups. Randomization will be performed by computer. Blinding of patients is not possible, but the observer will be blinded at eight weeks and six months.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years
* Grade II or III ankle sprains
* Presentation < 72 hours after the acute injury

Exclusion Criteria:

* Patients with a history of chronic instability
* Who had a fracture on X-ray investigation
* Other injuries or disabilities on the same limb
* Alcoholism, serious psychiatric and neurological illness
* Patients with bilaterally sprained ankles
* Patients with previous surgery on the lateral ankle ligaments
* Skin diseases where taping is not practicable
* Patients who are unable to give informed consent
* Patients who are unable to fill out questionnaires
* Neuromuscular disorders of the lower extremities
* Active rheumatoid arthritis
* Gait disturbances

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2010-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Karlsson score | up to 6 months FU
  The patients were asked to fill out a questionnaire regarding the function of the ankle joint. The score includes eight items based on a subjective evaluation of stability, pain, swelling and stiffness in relation to activities of everyday life, sports and recreational activities, running, stair climbing and working ability. The maximum score is 100 points.

SECONDARY OUTCOMES:
Return to work | up to 6 months FU
  Time to return to work Work at level / below level / no return to work
Return to sports | up to 6 months FU
  Time to return to sports Sports at level / below level /no return to sports
Pain VAS | up to 6 months FU
  VAS score 0-10: 0 = no pain, 10 = unbearable pain
Objective stability | up to 6 months FU
  Anterior Drawer Test (ADT). The patient sits on a bench with the legs hanging downwards. The knee joint is flexed and the foot held in 150 plantar flexion. First the healthy ankle is examined. Examination is performed according to van Dijk. 38 The examiner assigned one of the four predetermined numbers to each examined ankle joint, based on the estimated anterior displacement of the talus relative to the tibia.
  0 = 0-2mm, 1 = 3-5mm, 2 = 6-10mm and 3 = 11-15mm
Objective stability | up to 6 months FU
  DAAT. Because the manual ADT is of a subjective nature we measure the instability with the dynamic anterior ankle tester (DAAT). 39 The principle of the test is to apply a force impulse tot the calcaneus, within the muscle reflex time, and to measure anterior-posterior translation and mediolateral rotation. The highest and the lowest score were discarded and the mean of the three remaining scores counted as the result of the test.
Range of motion (ROM) | up to 6 months FU
  Degrees maximum dorsiflexion to plantarflexion
Recurrent inversion injury | up to 6 months FU
  Yes/no Number of sprains per month
Complications / adverse events | up to 6 months FU
  Any event leading to discontinuation of study participation and temporary or permanent physical damage due to the treatment under investigation (Local skin irritations (contact dermatitis and folliculitis), sensory deficit, stiffness, muscle atrophy). Use of not allowed painkillers is also an adverse event.
  * Yes / no
  * Total number of complications per patient and per group
Tegner activity level | up to 6 months FU
  Mean per group
EuroQol (EQ5D) | up to 6 months FU
  The EuroQol (EQ5D) is a health related quality of life instrument that provides a single index of an individual's quality of life. It consists of 5 dimensions resulting in 243 possible health states.
Costeffectiveness | up to 6 months FU
  Main objective of the economic evaluation is to assess the cost effectiveness and cost-utility of brace and tape therapy of acute lateral ankle ligament injury. The economic evaluation will be performed from a societal perspective, implying that both direct health care and direct non-health care costs, as well as indirect costs will be used as economic indicators. Firstly, relevant categories of resource utilisation were identified. Secondly, the volume of each category was measured and multiplied by the resource costs.
Compliance | up to 6 months FU
  How many full days did you not wear the (semi rigid / lace-up) brace? Tape compliance is always 100% (except in cases of complications / adverse events)
FAOS | up to 6 months FU
  FAOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport Rec), and foot and ankle-related Quality of Life (QOL). The last week is taken into consideration when answering the questionnaire. Standardized answer options are given (% Likert boxes) and each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. The result can be plotted as an outcome profile.

CONTACTS AND LOCATIONS:
Overall Officials: Eric EJ Raven, MD, Principal Investigator — Gelre Hospital
Locations (1):
- Gelre Hospitals, Apeldoorn, Netherlands